CLINICAL TRIAL: NCT01312285
Title: A Randomized, Double-blind, Placebo-controlled Evaluation of the Application of Magnetic Fields Using the Resonator Device for the Treatment of Osteoarthritis of the Hip: Pilot Study Protocol
Brief Title: Low Level Magnetic Fields for the Treatment of Osteoarthritis of the Hip
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: pico-tesla Magnetic Therapies, LLC (Industry)
Responsible Party: Allen S. Braswell CEO, pico-tesla Magnetic Therapies, LLC, CEO
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10276-01
Record Dates: First submitted 2011-01-10; First posted 2011-03-10 (Estimated); Last update posted 2011-05-30 (Estimated); Status verified 2011-05

CONDITIONS: Osteoarthritis of the Hip
Keywords: osteoarthritis; painful hips
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Device: Resonator device
- Resonator Device (Experimental)
  Interventions: Device: Resonator device

INTERVENTIONS:
Device: Resonator device — low level magnetic fields

SUMMARY:
The purpose of this study is to see if using a device called the Resonator, that puts out very low level electromagnetic fields will help symptoms of painful hip(s)

DETAILED DESCRIPTION:
The purpose of this pilot study is to assess the efficacy of the Resonator™ device, manufactured by Pico-Tesla, the MAGNECEUTICAL® company (the Sponsor), as an adjunctive therapy to reducing pain and improving function for individuals with osteoarthritis of the hip.

ELIGIBILITY:
Inclusion Criteria:

* > Diagnosis of osteoarthritis of the hip for at least one hip (right or left hip, or both hips) determined by satisfaction of BOTH of the following (as outlined in the STUDY TEST BATTERY section above):

  * the American College of Rheumatology (ACR) Classification Criteria for osteoarthritis of the hip, AND
  * Rating of current Degree of Pain in the hip on the 0-100 Visual Analog Scale of 40 or greater.

N.B.: If both hips satisfy both of the above criteria for diagnosis of osteoarthritis of the hip, the hip with the highest VAS pain rating will be selected for evaluation in this study. That is, only one hip per subject will be evaluated in this study.

* Hip pain was present on most days of the prior three months.
* Subject is ambulatory.
* Subject's use of pain relief medication(s) has been stable over the past 30 days, and the subject is willing and able to maintain this existing use of pain relief medication(s) as his or her sole pain relief medication use, as needed, throughout study participation.
* Subject has been on current non-pain relief medication regimen (for any indication or condition such as hypertension, pulmonary disease or cardiac disease), unchanged, or on no current non-pain relief medication regimen, for at least 30 days prior to study enrollment, and is willing and able to maintain his or her regular non-pain relief medication regimen, unchanged, throughout the course of his or her study participation unless the subject's physician states that a medication change is needed for the subject's safety and well-being, in which case the subject agrees to inform the study PI of the change(s) made ,.
* Willing and able to abstain from partaking in other/new treatments (other than the study procedures) to improve osteoarthritis of the hip pain and other symptoms during the course of participation in the study. Such treatments include new medications, dietary/herbal supplements/ minerals, weight loss programs, water or other new exercise programs, physical therapy, occupational therapy, surgical procedures, and alternative therapies such as acupuncture, massage, or hypnotherapy.
* Adequate contraceptive measures for female subjects. > 18 years of age or older.
* Male or female.

Exclusion Criteria:

* > Neither the right nor the left hip satisfies BOTH of the following criteria for a diagnosis of osteoarthritis of the hip (as outlined in the STUDY TEST BATTERY section):

  * the American College of Rheumatology (ACR) Classification Criteria for osteoarthritis of the hip, AND
  * Rating of current Degree of Pain in the hip on the 0-100 Visual Analog Scale of 40 or greater.

    * Hip pain was not present on most days of the prior three months.
    * Subject is non-ambulatory.
    * Any factors that might prevent the subject from completing a full course of therapy with the Resonator™ device, or from attending any of the scheduled study visits during the planned study duration, or from completing any of the study measures.
    * Any other significant comorbidities that might impact the ability to evaluate the subject's satisfaction of the American College of Rheumatology Classification Criteria for osteoarthritis of the hip, or for the subject to complete any of the study assessment tools.
    * Subject's use of pain relief medication(s) has not been stable over the past 30 days and/or the subject is not willing and/or unable to maintain this existing use of pain relief medication(s) as his or her sole pain relief medication use, as needed, throughout study participation.
    * Not willing and/or unable to abstain from partaking in new treatments (other than the study procedures) to improve osteoarthritis of the hip pain and other symptoms during the course of participation in the study. Such treatments include new medications, dietary/herbal supplements/minerals, weight loss programs, water or other new exercise programs, physical therapy, occupational therapy, surgical procedures, and alternative therapies such as acupuncture, massage, or hypnotherapy.
    * An intra-articular hip injection (with any corticosteroid, hyaluronic acid preparation or other) within the prior three months.
    * Known inflammatory rheumatic disease.
    * Epilepsy/history of seizures/taking medication for epilepsy.
    * HIV and other autoimmune disorders.
    * Active cancer or treatment for cancer within last 6 months.
    * Confirmed active infection(s).
    * Signs of clinically important active inflammation of the hip joint including redness, warmth, swelling and/or a large, bulging effusion with the loss of normal contour.
    * Acute inflammation or ischaemic necrosis.
    * Inflammatory arthropathy of the hip.
    * Inflammatory system diseases that could interfere with the evaluation of the study procedure.
    * Hip arthropathy due to diabetes mellitus.
    * Charcot's joint.
    * Villous synovitis.
    * Chondromatosis of the synovium.
    * Rapid destructive hip.
    * History of crystalline arthropathy or inflammatory arthritis, neuropathic arthropathy.
    * Secondary osteoarthritis of the study hip joint including, but not limited to, septic arthritis, inflammatory joint disease, gout, Paget's disease of bone, articular fracture, major dysplasias or congenital abnormality, ochronosis, acromegaly, hemochromatosis, Wilson's disease, avascular necrosis, or primary osteochondromatosis.
    * History of acute inflammatory arthritis or pseudogout of the study hip.
    * History of ECT.
    * Uncontrolled hypertension.
    * Advanced pulmonary disease.
    * Unstable cardiac disease, such as any history of cardiac arrhythmias (including atrial fibrillation, ventricular fibrillation, or irregular atrial-ventricular conduction time), or any incidences of congestive heart failure, or myocardial infarction, within the last six months.
    * Prosthetics or implants comprised of ferrous metals.
    * History of surgery, including arthroscopy, or major trauma to the study hip joint in the prior six months.
    * Endoprothetic replacement of study hip joint.
    * Pacemakers, vagus nerve stimulators, or other functional electrical stimulators such as those commonly used for pain.
    * Reported consumption of more than 21 alcoholic drinks per week.
    * Pregnant, breast feeding, or planning pregnancy prior to the end of participation.
    * Current or past history of major psychiatric disturbance (e.g., schizophrenia, bipolar disorder, substance abuse). However, subjects with a history of adequately treated depression or anxiety disorders will not be excluded. Anti-depressant drug therapy must be stable for at least 4 weeks prior to study entry and must remain stable throughout study duration.
    * Developmental disability or other cognitive impairment that would in the judgment of the PI impair adequate comprehension of the informed consent form or complete any of the study-related activities.
    * Worker's compensation (current or pending), current receipt of disability or present /past litigation for monetary compensation pertaining to the subject's osteoarthritis of the hip condition.
    * Participation in investigational drug or medical device research within 30 days of enrollment in this current pilot study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-03 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
The mean change from baseline to study endpoint in the 3-recording average of the subject's Daily Pain Rating on the 0-100 VAS for the study hip recorded each morning upon waking and prior to consuming any pain medication for the day. | 14 days

SECONDARY OUTCOMES:
Daily morning recordings of pain intensity ratings for the study hip on the 0-100 VAS | 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- Innovative Research, Clearwater, Florida, United States